CLINICAL TRIAL: NCT00834769
Title: Chronic Pain After Thoracotomy, an Incidence Study in a Single Surgical Center
Status: Completed | Type: Observational
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Other Study IDs: 2008/30
Record Dates: First submitted 2009-02-02; First posted 2009-02-03 (Estimated); Last update posted 2016-09-23 (Estimated); Status verified 2016-09

CONDITIONS: Thoracotomy; Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Investigation of chronic pain frequency after thoracotomy for lung cancer. Risk factors for development of chronic pain are investigated. Questionnaire survey.

ELIGIBILITY:
Inclusion Criteria:

* thoracotomized patients

Exclusion Criteria:

* mental incapacity,
* poor understanding of French,
* pre-existing chronic pain before surgery,
* redo-surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: thoracotomized patients
Sampling Method: Non-Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2008-12; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Pain and pain score | one year postoperative

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital Foch, Suresnes, France